CLINICAL TRIAL: NCT06020430
Title: Omitting CTV Radiotherapy for Locally Advanced Non Small Cell Lung Cancer Responded to Immunotherapy and Radiotherapy
Brief Title: Omitting CTV for Locally Advanced NSCLC Responded to Immunotherapy and Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hubei Cancer Hospital (Other)
Responsible Party: Principal Investigator, HAN GUANG, Director of the department of Radiotherapy Oncology, Hubei Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OMCTV-HC-001
Record Dates: First submitted 2023-08-28; First posted 2023-08-31 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Non Small Cell Lung Cancer; Locally Advanced; Radiotherapy; Immunotherapy
Keywords: omitting CTV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTV-omitted (Experimental): CTV was omitted for the radical radiotherapy for locally advanced NSCLC who responded to induction therapy with immunotherapy and chemotherapy.
  Interventions: Radiation: CTV omitted or delineated
- CTV-delineated (Active Comparator): CTV was delineated for the radical radiotherapy for locally advanced NSCLC who responded to induction therapy with immunotherapy and chemotherapy.
  Interventions: Radiation: CTV omitted or delineated

INTERVENTIONS:
Radiation: CTV omitted or delineated — Patients who responded to the induction therapy (immunotherapy and chemotherapy) were randomly (1:1) assigned into CTV-omitted radical radiotherapy group or CTV-delineated radiotherapy group.

SUMMARY:
Radical radiotherapy is critical for locally advanced non small cell lung cancer(NSCLC ). Our previous sturdy indicated that patients who received induction immunotherapy and subsequent radiotherapy suffered higher proportion of pneumonitis.Grade 2 or more pneumonitis patients have worse prognosis. It is urged to optimize the radiotherapy dose and target volume for patients treated with immunotherapy and radiotherapy. According to retrospective and prospective studies, omitting CTV radiation is feasible for patients undergoing concurrent radio-chemotherapy for locally advanced NSCLC. It is postulated that omitting CTV radiation for patients responded to induction therapy with immunotherapy and chemotherapy will have less pneumonitis without sacrificing the local control rate. Omitting CTV may also retain better immune function which will facilitate the immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed non-small cell lung cancer;
2. stage IIIA or IIIB or IIIC according to the 8th edition of the TNM cancer staging system of the American Joint Committee on Cancer (AJCC) and Union for International Cancer Control（UICC);
3. inoperable or refuses surgery after induction therapy with immunotherapy and chemoradiotherapy;
4. After ≥2 cycles of induction chemotherapy combined with immunotherapy, the efficacy was CR, PR or SD (with a decreasing trend);
5. performance status 0-1;
6. measurable or evaluable lesions;
7. Survival expectancy is not less than 6 months;
8. adequate cardiac, pulmonary, renal, and hepatic and bone marrow function

Exclusion Criteria:

1. tumor progress after induction with immunothearoy and chemotherapy
2. EGFR, ALK, or ROS1 mutation;
3. Previous thoracic radiotherapy;
4. grade 2 or more immune-related adverse events after induction immunotherapy
5. Previous malignancies (except stage I non-melanic skin cancer or cervical carcinoma in situ);
6. Pregnant or lactating women
7. undergoing other clinical trials;
8. Have serious comorbidities, including myocardial infarction, severe arrhythmia, severe cerebrovascular disease, ulcer disease, psychosis and uncontrollable diabetes;
9. Patients with HIV positive and undergoing antiviral therapy;
10. Active tuberculosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2026-02-08 (Estimated); Study Completion 2027-10-08 (Estimated)

PRIMARY OUTCOMES:
grade 2 or more pneumonitis | up to 6 months

SECONDARY OUTCOMES:
local/regional control rate | up to 12 months
Progress free survival | up to 12 months
grade 3 or more pneumonitis | up to 6 months
grade 3 or more esophagitis | up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hubei Cancer Hospital, Wuhan, Hubei, China